CLINICAL TRIAL: NCT05970432
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial Evaluating the Efficacy and Safety of TQH2722 Injection in Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Clinical Study of TQH2722 Injection in the Treatment of Moderate to Severe Atopic Dermatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQH2722-II-01
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TQH2722 injection 300mg-150mg (Experimental): Participants received subcutaneous injection of 300 mg TQH2722 injection + 600 mg placebo on day 1, followed by subcutaneous injection of 150 mg TQH2722 injection + 300 mg placebo on days 15, 29, 43, 57, 71, 85, 99.
  Interventions: Drug: TQH2722 injection 300mg-150mg
- TQH2722 injection 600mg-300mg (Experimental): Participants received subcutaneous injection of 600 mg TQH2722 injection + 300 mg placebo on day 1, followed by subcutaneous injection of 300 mg TQH2722 injection + 150 mg placebo on days 15, 29, 43, 57, 71, 85, 99.
  Interventions: Drug: TQH2722 injection 600mg-300mg
- TQH2722 injection 900mg-450mg (Experimental): Participants received subcutaneous injection of 900 mg TQH2722 injection on day 1, followed by subcutaneous injection of 450 mg TQH2722 injection on days 15, 29, 43, 57, 71, 85, 99.
  Interventions: Drug: TQH2722 injection 900mg-450mg
- TQH2722 injection matching Placebo (Placebo Comparator): Subjects received 900mg placebo injection subcutaneously on day 1, followed by 450mg placebo injection on days 15, 29, 43, 57, 71, 85, 99.
  Interventions: Drug: TQH2722 injection matching Placebo

INTERVENTIONS:
Drug: TQH2722 injection 300mg-150mg — TQH2722 injection is a fully human monoclonal antibody that interfering with the signal cascade.
  Arms: TQH2722 injection 300mg-150mg
Drug: TQH2722 injection 600mg-300mg — TQH2722 injection is a fully human monoclonal antibody that thereby interfering with the signal cascade.
  Arms: TQH2722 injection 600mg-300mg
Drug: TQH2722 injection 900mg-450mg — TQH2722 injection is a fully human monoclonal antibody that thereby interfering with the signal cascade.
  Arms: TQH2722 injection 900mg-450mg
Drug: TQH2722 injection matching Placebo — Placebo without active substance.
  Arms: TQH2722 injection matching Placebo

SUMMARY:
This phase II clinical trials is multicenter, randomized, double-blind, placebo-controlled to assess the effectiveness and safety of TQH2722 injection in the treatment of subjects with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 (when signing informed consent), regardless of gender;
* Meets 2014 American Academy of Dermatology (AAD) criteria with diagnosis of atopic dermatitis (AD); In addition, history of AD prior to screening ≥ 6 months; Eczema was previously diagnosed but met the 2014 AAD criteria and can still be enrolled.
* Patients with moderate to severe AD at screening and baseline visit (shall meet all 3 criteria as follows):

  1. total area of AD lesions≥ 10% BSA;
  2. IGA ≥3 points;
  3. EASI ≥ 16 points;
* Baseline peak pruritus NRS ≥4 (The average peak pruritus intensity score in baseline peak pruritus NRS will be calculated based on the average of the peak pruritus intensity NRS score (daily score range 0-10) for each day during the 7 days prior to randomization. A minimum of 4 days out of 7 days of scoring is required to calculate the baseline average score. If the patient's reporting days are less than 4 days in the 7 days prior to the planned randomization date, randomization should be postponed until the requirements are met, but not beyond the maximum period of 14 days for screening);
* 6 months prior to the screening period, insufficient response to stable (≥1 month) topical corticosteroids (TCS) or calcineurin inhibitors (TCI) (insufficient response defined as at least 28 days even if the daily regimen of moderate-high potency TCS (± topical TCI, if applicable) is at least 28 days, or to the maximum recommended course of treatment (eg, ultra-potent TCS - 14 days) in the product prescribing information (whichever is shorter), Failure to achieve or maintain disease remission or low disease activity (equivalent to IGA 0 [=none]-2 [=mild]). or patients who have received a record of systemic treatment (adequate dose, adequate course) of AD in the past 6 months are also considered to have insufficient response to topical drug therapy, and may be selected for trial after appropriate drug elution and approval by the sponsor);
* Before the first dose, subjects must have continuously used the emollient twice a day for at least 1 week and maintained throughout the trial (Note: the emollient is provided by the sponsor);
* Be able to read and understand, and be willing to sign informed consent forms;
* Willingness and compliance with research visits and related procedures;
* Female participants of childbearing age should agree that contraception (e.g., intrauterine devices, pills, or condoms) must be used during the study period and for 6 months after the end of the study; Negative serum pregnancy test within 7 days prior to first dose and must be a non-lactating subject; Male subjects should agree that contraception must be used during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

* Participants who received the following treatments within the following limited time prior to randomization:

  1. Have used any of the following treatments within 4 weeks or the investigator believes that the following treatments may be required: immunosuppressants/immunomodulatory drugs (eg, systemic glucocorticosteroids, cyclosporine, mycophenolate mofetil, interferon γ (IFN-γ), azathioprine, and methotrexate); AD phototherapy;
  2. Oral Janus Kinase (JAK) inhibitors (including but not limited to upadacitinib) used within 2 weeks;
  3. Received systemic traditional Chinese medicine (TCM) treatment within 4 weeks; or within 1 week, topical TCM;
  4. Treated with leukotriene inhibitors within 4 weeks;
  5. Treated with topical preparations of TCS or TCI or phosphodiesterase 4 (PDE⁃4) inhibitors within 2 weeks;
  6. Treatment with the following biologics: any cell depleting agent, including but not limited to rituximab: within 6 months or until the lymphocyte count returns to normal, whichever is longer; Other biologics: 5 half-lives (if half-life known) or 12 weeks (whichever is longer); Within 4 weeks, receive regular phototherapy (including but not limited to narrow-spectrum UVB, psoralen longwave ultraviolet therapy, etc.) or use artificial sunbathing sheds/rooms;
  7. Within 12 weeks, receive live (attenuated) vaccine;
  8. Chronic active or acute infection requiring systemic treatment with antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks, or superficial skin infection within 1 week prior to baseline visit. After the infection resolves, screening can be renewed;
  9. Antihistamines (including oral, nasal, and topical preparations) within 1 week;
* Abnormal physical examination results during screening or any of the following laboratory tests:

  1. Hemoglobin< 110 g/L
  2. White blood cell (WBC) < 3.5 x 10^9/L
  3. Platelet count < 125 x 10^9/L
  4. Neutrophils< 1.75 x 10^9/L • Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >1.5 x upper limit of normal (ULN)
  5. Total bilirubin > 1.5 x ULN (except indirect bilirubin elevation secondary to Gilbert syndrome)
  6. Creatinine > 1.5 x ULN
  7. Creatine phosphokinase (CPK) > 2 x ULN
* There are cutaneous comorbidities that may interfere with the study assessment, including but not limited to scabies, seborrheic dermatitis, cutaneous T-cell lymphoma, psoriasis, etc
* Concomitant other serious medical conditions that, at the discretion of the investigator, may adversely affect participants' participation in this study, including, but not limited to: short life expectancy, history of uncontrolled diabetes (HbA1c ≥ 9%), cardiovascular disease (eg, grade III or IV heart failure, graded according to the New York Heart Association), severe kidney disease (eg, patients on dialysis), hepatobiliary disease (e.g., Child-Pugh class B or C), neurological disease (e.g., demyelinating disease), Patients with important active autoimmune diseases (eg, lupus, inflammatory bowel disease, rheumatoid arthritis, etc.), as well as other severe endocrine, gastrointestinal, metabolic, pulmonary, or lymphatic diseases.
* Have a history of known or suspected immunosuppression, including invasive opportunistic infections (e.g., histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, and aspergillosis), even if the infection has resolved; or unusual frequent, recurrent, or long-term infections (at the investigator's discretion);
* Subjects with any type of active malignancy or a history of malignancy (except cervical cancer or non-metastatic cutaneous squamous cell carcinoma, basal cell carcinoma and papillary thyroid carcinoma) that has been cured for more than 5 years prior to the screening period;
* Computed Tomography (CT) of the chest shows active or occult tuberculosis or a history of contact with an open tuberculosis (TB) subject within the past 6 months. If the laboratory T cell spot test for tuberculosis infection test (or other tuberculosis diagnostic test) is positive, its activity is judged in combination with the medical history, clinical manifestations, etc., and the investigator determines whether it can be enrolled;
* Active hepatitis during the screening period, or positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis B core antibody (HBcAb);
* History of human immunodeficiency virus (HIV) infection, or positive HIV serological results at screening, and positive antibodies to treponema pallidum during screening
* Positive for treponemal pallidum antibodies during screening
* Parasitic infection related to any of the following is excluded:

  1. Routine inspection of worm eggs during the screening period;
  2. History of parasitic infection within 6 months prior to the screening period, except for cured trichomoniasis;
* Have participated in clinical trials of other drugs or medical devices within 12 weeks prior to screening
* During the period of participation in this study, participants had planned surgical procedures
* Pregnant or lactating women
* People who are alcoholic, drug addicts, and known drug dependents
* In the judgment of the investigator or sponsoring medical auditor, it is believed that there are any medical or psychiatric symptoms that put the subject at risk, interfere with participation in the study, or interfere with the interpretation of the results of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Eczema area and severity (EASI)-75 (≥75% improvement from baseline). | Up to 16 weeks.
  Proportion of participants with eczema area and severity (EASI)-75 (≥75% improvement from baseline) at week 16.

SECONDARY OUTCOMES:
Investigator's general assessment (IGA) | Up to 16 weeks.
  Proportion of subjects with, the investigator's overall assessment (IGA) of 0 or 1 (6-point in total) at week 16.
Eczema area and severity (EASI)-90 (≥90% improvement from baseline). | Up to 16 weeks.
  Proportion of participants with EASI-90 at week 16.
Eczema area and severity (EASI) | Up to 16 weeks.
  Percentage change in EASI score from baseline to week 16;
Change in investigator's general assessment (IGA) | Up to 16 weeks.
  Change (or percentage change) in IGA score from baseline to week 16;
Body surface area (%BSA) | Up to 16 weeks.
  %BSA change from baseline to week 16
Treatment Emergent Adverse Events (TEAE) | Up to 20 weeks.
  Incidence of TEAE from baseline to week 20 determined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTC AE) V5.0.
Incidence of anti-drug antibodies (ADAs) | Up to 24 weeks.
  The incidence of anti-drug antibodies (ADAs) of subjects and their titer, the incidence of neutralizing antibodies (Nab). If the subject is tested positive for ADA, a neutralizing antibody is added in the test.
Incidence of neutralizing antibodies | Up to 24 weeks.
  If the subject is tested positive for ADA, a neutralizing antibody is added.
Peak Itch numerical rating scale (NRS) | Up to 16 weeks.
  Peak Itch NRS changes from baseline to week 16. The total score is 10, with higher scores indicating more severe pruritus.
Dermatology Life Quality Index (DLQI) scores | Up to 16 weeks.
  DLQI scores change from baseline to week 16, the scores are rated as None, Not Relevant, and 0-3, with higher values representing more serious disease.

CONTACTS AND LOCATIONS:
Locations (32):
- China (32):
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Dermatology Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Affiliated Hospital of Hebei Engineering University, Handan, Hebei
  - The Forth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The second affiliated hospital of harbin medical university, Harbin, Heilongjiang
  - Puyang District Hospital of Anyang City, Anyang, Henan
  - The First People's Hospital of Nanyang, Nanyang, Henan
  - People's Hospital of Henan province, Zhengzhou, Henan
  - Shiyan Renmin Hospital, Shiyan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The third xiangya hospital of central south university, Changsha, Hunan
  - Qian-jin Lu, Nanjing, Jiangsu
  - Affiliated Hospital of Jiujiang University, Jiujiang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Panjin Liaoyou Gem Flower Hospital, Panjin, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Air Force Medical University, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shengli Oil Field Central Hospital, Dongying, Shandong
  - Shandong First Medical University Affiliated Dermatology Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Hospital Of Qingdao University, Qingdao, Shandong
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Uygur Autonomous Region People's Hospital, Ürümqi, Xinjiang Uygur Autonomous Region
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First People's Hospital of Wenling, Wenling, Zhejiang